CLINICAL TRIAL: NCT05668195
Title: Research and Promotion of Systematic Aerobic Exercise and Intelligent Monitoring System in Executive Skill Training for School-aged Children With Attention Deficit Hyperactivity Disorder
Brief Title: Systematic Aerobics and Intelligent Monitoring System in Executive Skill Training for School-aged Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Li (Other)
Collaborators: Southwest University, China (Unknown)
Responsible Party: Sponsor-Investigator, Chen Li, Associate Professor, Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEIMS
Record Dates: First submitted 2022-12-09; First posted 2022-12-29 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: ADHD
Keywords: ADHD, Executive Skill Training, Aerobic Exercise
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The children in the group are randomly divided into a test group and a control group, and further divided into 4 groups according to whether they were also treated with medication (methylphenidate) or not. Children receiving methylphenidate are required to be titrated to a stable dose before training, and those who did not change medication, stop medication, or adjust dose during training are included in the analysis. The test group receive systematic aerobic exercise and intelligent monitoring system in executive skill training, the control group receive systematic executive skill training, for 13 weeks. The research team, together with other teams, has initially developed a set of closed-loop training and is further exploring it in training.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise group (Experimental): The patients aged 6-12 with a diagnose of ADHD of this group receive systematic aerobic exercise and intelligent monitoring system in executive skill training for 13 weeks, including those taking methylphenidate or not.
  Interventions: Procedure: systematic aerobic exercise and intelligent monitoring system in executive skill training; Procedure: executive skill training
- executive skill training group (Active Comparator): The patients aged 6-12 with a diagnose of ADHD of this group receive executive skill training for 13 weeks, including those taking methylphenidate or not.
  Interventions: Procedure: executive skill training

INTERVENTIONS:
Procedure: systematic aerobic exercise and intelligent monitoring system in executive skill training — This is a closed-loop training initially developed by the research team in conjunction with other teams, adding a systematic aerobic exercise and intelligent monitoring system to the typical executive skill training, and is being further explored in training.
  Arms: aerobic exercise group
Procedure: executive skill training — The training program, based on Dawson and Guare's (2010) training of executive skills for children, aimed to improve the everyday performance of executive skills among children with ADHD. Qian Y and her team added some culturally adapted information, following the theory of cognitive behavioral therapy, to ensure that the concepts were acceptable to Chinese children.

SUMMARY:
Around 7.2% of children around the world are suffering from Attention Deficit Hyperactivity Disorder (ADHD). Systematic executive skill training for children is currently recognized as one of the main programs for psychosocial behavioral interventions in ADHD, but the theoretical basis for the 1 hour "play class" component of the 3 hours per week children's classroom is insufficient. We have developed a closed-loop moderate-intensity aerobic training system, which is combined with an intelligent monitoring system, to further standardize and improve the treatment and management of ADHD intervention. The intelligent monitoring system in this study includes physiological intelligent monitoring (heart rate data) and psychological and behavioral intelligent monitoring (based on the computerized "adaptive" executive function testing procedures and clinical questionnaire scale). 200 subjects aged 6-12 years with a diagnosis of ADHD based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria are randomly assigned into two groups to receive executive skill training and systematic aerobic exercise and intelligent monitoring system, or systematic executive skill training for 13 weeks. Symptoms severity is assessed by Vanderbilt Assessment Scales at weeks 0, 6, and 13. Subjects' executive function is assessed using executive function tests before and after training, parental depression/anxiety assessment, family environment assessment, and monitoring of heart rate during exercise are also included. All the other sociodemographic data are assessed. This study will investigate the effects of systematic aerobic exercise and intelligent monitoring system in executive skill training on the promotion of cold executive functions such as responsiveness, flexibility, and inhibition and hot executive functions such as reward mechanisms in children, and their effects on children with ADHD and their families.

DETAILED DESCRIPTION:
1. Procedures. The children in the group are randomly divided into a test group and a control group, and further divided into 4 groups according to whether they were also treated with medication (methylphenidate) or not. Children receiving methylphenidate are required to be titrated to a stable dose before training, and those who did not change medication, stop medication, or adjust dose during training are included in the analysis. The children will be trained for 13 weeks, and the children with ADHD will be evaluated for symptoms and functions, parenting stress, and family environment at training weeks 0, 6, and 13, respectively; the children will be tested for executive function at training weeks 0 and 13; and the children with ADHD will be monitored for basic vital indicators.
2. Demographic questionnaire and clinical data. The demographic questionnaire is completed by the child's primary caregiver, detailing child's name, gender, date of birth, height, weight, blood pressure, heart rate. Clinical data will be ascertained from the medical records, including information about DSM-5 diagnosis, disease classification, current treatment, and comorbid conditions.
3. Sample size. This study is a randomized controlled trial. Intervention group receives executive skill training and systematic aerobic exercise and intelligent monitoring system, control group receives systematic executive skill training. The primary outcome index is changes in ADHD symptoms evaluated by Vanderbilt Assessment Scales and changes in executive functions evaluated by executive function tests such as Stop-Signal task, GO/NO-GO task reflecting response control, Simon task reflecting conflict control, Dimensional Change Card Sorting (DCCS) task reflecting cognitive flexibility, and N-Back task reflecting working memory. Self-rating depression scale, self-rating anxiety scale are used to assess parental emotions, family environment scale-Chinese version is used to assess family environment. The child wears a heart rate band to monitor heart rate changes during exercise and the data is collected and analyzed in the background. Since this study is pioneering, the investigators artificially set the sample size at 200.
4. Statistical analysis. All the data are analyzed using SPSS 25.0. The normality of variables are assessed by Kolmogorov Smirnov test. Comparison of parametric and nonparametric variables between groups are examined by F test and Kruskal-Wallis test, respectively. Paired t-test and Wilcoxon signed-rank test are used to investigate within-group differences. Confounding factors are adjusted by the analysis of covariance.
5. Ethical matters and data protection. The patients participated in the study will sign the informed consent (obtained from the guardian). And this study was approved by the local ethics committee. Patient's name will be abbreviated and the research data will be assigned a code then to provide to the researcher. The authorization from parents on the patient's health information remains valid until the study is completed. After that, researchers will delete private information from the study record.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of ADHD according to DSM-5
* Aged 6-12 years
* Children receiving methylphenidate are required to be titrated to a stable dose before training, and those who did not change medication, stop medication, or adjust dose during training are included in the analysis

Exclusion Criteria:

* IQ≤80
* Inconsistent or changing dose of methylphenidate during the participation period
* Suffering from organic lesions of nervous system now or in the past
* Suffering from epilepsy, autism spectrum disorder and other severe neurodevelopmental behavioral disorders now or in the past
* Not suitable for medium to high intensity aerobic training

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes in ADHD clinical symptoms-Estimated by Chinese version of Vanderbilt parent/teacher diagnostic scale | at weeks 0 for the children with first diagnosis of ADHD
  The Vanderbilt parent/teacher diagnostic scale is designed to measure the severity of ADHD symptoms for children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 49-56/36-43 are performance measures. The symptom measures in the scale, scored 0 to 3. A positive response in symptom assessment part is a 2 or 3 (often, very often). The performance measures in the scale, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  The scoring standard: Must score a 2 or 3 on 6 out of 9 items on questions 1-9(Predominantly Inattentive subtype)/10-18(Predominantly Hyperactive/Impulsive subtype)/both 1-9 and 10-18(ADHD Combined Inattention/Hyperactivity) AND Score a 4 or 5 on any of the Performance questions 49-56(parent)/36-43(teacher). The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Estimated by Chinese version of Vanderbilt parent/teacher follow-up scale | at weeks 0, 6 and 13
  The Vanderbilt parent/teacher follow-up scale is designed to track treatment effect over time for ADHD children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 19-26 are performance measures. The symptom measures in the scale, scored 0 to 3 (Never, Occasionally, Often, Very Often). The performance measures in the scale, scored 1 to 5 (Excellent, Above Average, Average, Somewhat of a Problem, Performance Problematic).
  The scoring standard: 1) Calculate Total Symptom Score for questions 1-18. 2) Calculate Average Performance Score for questions 19-26. The higher scores mean a worse outcome.
False alarms of GO/NO-GO task | at weeks 0 and 13
  GO/NO-GO task reflects response inhibition. Subjects are required to press a button when a certain stimulus appeared on the screen (e.g., a circle) and not when some other stimulus appeared (e.g., a triangle), with the majority of stimuli requiring a button (≥75%) and a small percentage of stimuli not requiring a button (≤25%). The false alarms are the numbers of stimuli to which subjects responded incorrectly that did not require a response.
The correct rate of GO/NO-GO task | at weeks 0 and 13
  GO/NO-GO task reflects response inhibition. Subjects are required to press a button when a certain stimulus appeared on the screen (e.g., a circle) and not when some other stimulus appeared (e.g., a triangle), with the majority of stimuli requiring a button (≥75%) and a small percentage of stimuli not requiring a button (≤25%). We will calculate the correct rate.
The correct rate of Stop-signal task | at weeks 0 and 13
  Similar to GO/NO-GO task, Stop-signal task also reflects response inhibition. The "GO" signal presents every time, but in a few instances the "GO" signal is followed by a "Stop" signal, when the subject was asked not to press the button. The majority of stimuli (≥75%) require to press a button, while the "GO" signal followed by a "Stop" signal is ≤25%. We will calculate the correct rate.
The correct rate of Simon task | at weeks 0 and 13
  Simon task reflects interference control. When subjects see stimulus A, press the left button (L); when they see stimulus B, press the right button (R). Stimuli A and B may appear in different directions. We will calculate the correct rate.
The number of correct switches of DCCS task | at weeks 0 and 13
  DCCS task reflects cognitive flexibility. Subjects are presented with a set of stimulus pictures with different dimensions (such as shape, number and color) and test pictures that can be matched with different stimulus pictures in different dimensions. Subjects need to classify the current stimulus according to different rules. When the rules change, they need to adjust their reactions as soon as possible and change the classification way. The number of correct switches refers to the number of times the subject continuously makes the correct response when the classification rule is changed.
The correct rate of DCCS task | at weeks 0 and 13
  DCCS task reflects cognitive flexibility. Subjects are presented with a set of stimulus pictures with different dimensions (such as shape, number and color) and test pictures that can be matched with different stimulus pictures in different dimensions. Subjects need to classify the current stimulus according to different rules. When the rules change, they need to adjust their reactions as soon as possible and change the classification way. We will calculate the correct rate.
The hit rate and the false alarm rate of N-back task | at weeks 0 and 13
  N-back task reflects working memory. The subjects are presented with a series of stimuli and asked to compare the current stimulus with the Nth stimulus backwards. If the two stimuli are the same, it is the target; if they are different, it is the non-target. The hit rate means that the subject responds correctly to the target, and the false alarm rate means that the subject responds incorrectly to the non-target.

SECONDARY OUTCOMES:
The changes of parental mood-Estimated by Self-rating depression scale (SDS) | at weeks 0, 6 and 13
  The Self-Rating Depression Scale (SDS) consists of 20 items with a Likert type scale after each item. The scores for each item range from 1 to 4 and the SDS ranges from a raw score of 20 to a raw score of 80. Some items are reverse scored (i.e., they go from 4 down to 1). SDS scores are classified as normal (<50), mild depression (50 to 59), moderate to marked major depression (60 to 69), and severe to extreme major depression (>70). The raw score can be converted to an SDS Index score by multiplying the raw score times 1.25.
The changes of parental mood-Estimated by Self-rating anxiety scale (SAS) | at weeks 0, 6 and 13
  The SAS groups anxiety manifestations into cognitive, autonomic, motor, and central nervous system symptoms. Each of the 20 items is answered on a four-point Likert scale ranging from 1 to 4:1 - A little of the time, 2 - Some of the time, 3 - A good part of the time, 4 - Most of the time. A person's score is calculated by adding up all the values selected. Higher scores indicate greater levels of anxiety. According to Zung, the total raw scores are converted to an anxiety index number using a conversion chart. The anxiety index numbers are interpreted as follows: Less than 45: Normal range, 45-59: Mild to moderate anxiety levels, 60-74: Marked to severe anxiety levels, 75-80: Extreme anxiety levels.
The changes of family environment-Estimated by Family environment scale-Chinese version (FES-CV) | at weeks 0, 6 and 13
  The Family Environment Scale is a 90 item measure that evaluates the social environment of the family unit. Three forms are available: the Real Form (Form R), which measures the family environment as it is; the Ideal Form (Form I) which measures the family environment as it would be in a perfect situation; and the Expected Form (Form E), which measures the family environment as it will probably be in new situations. The FES is composed of ten subscales that measure the underlying dimensions of Family Relationship, Personal Growth and System Maintenance and Change.
The changes in heart rate | during the class of aerobic exercise, about 40min per class, once a week, 13weeks
  Heart rate (or pulse rate) is the frequency of the heartbeat measured by the number of contractions (beats) of the heart per minute (bpm). When the children are doing aerobic exercise, we monitor the changes of heart rate and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University; yu T Li, MS, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Growth, Development and Mental health of Children and Adolescence Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Background] Wolraich ML, Hagan JF Jr, Allan C, Chan E, Davison D, Earls M, Evans SW, Flinn SK, Froehlich T, Frost J, Holbrook JR, Lehmann CU, Lessin HR, Okechukwu K, Pierce KL, Winner JD, Zurhellen W; SUBCOMMITTEE ON CHILDREN AND ADOLESCENTS WITH ATTENTION-DEFICIT/HYPERACTIVE DISORDER. Clinical Practice Guideline for the Diagnosis, Evaluation, and Treatment of Attention-Deficit/Hyperactivity Disorder in Children and Adolescents. Pediatrics. 2019 Oct;144(4):e20192528. doi: 10.1542/peds.2019-2528. PMID 31570648
- [Background] Brown TE. ADD/ADHD and Impaired Executive Function in Clinical Practice. Curr Psychiatry Rep. 2008 Oct;10(5):407-11. doi: 10.1007/s11920-008-0065-7. PMID 18803914
- [Background] Brown TE, Holdnack J, Saylor K, Adler L, Spencer T, Williams DW, Padival AK, Schuh K, Trzepacz PT, Kelsey D. Effect of atomoxetine on executive function impairments in adults with ADHD. J Atten Disord. 2011 Feb;15(2):130-8. doi: 10.1177/1087054709356165. Epub 2009 Dec 21. PMID 20026871
- [Background] Qian Y, Chen M, Shuai L, Cao QJ, Yang L, Wang YF. Effect of an Ecological Executive Skill Training Program for School-aged Children with Attention Deficit Hyperactivity Disorder: A Randomized Controlled Clinical Trial. Chin Med J (Engl). 2017 Jul 5;130(13):1513-1520. doi: 10.4103/0366-6999.208236. PMID 28639564
- [Background] Diamond A, Lee K. Interventions shown to aid executive function development in children 4 to 12 years old. Science. 2011 Aug 19;333(6045):959-64. doi: 10.1126/science.1204529. PMID 21852486
- [Background] Liang X, Li R, Wong SHS, Sum RKW, Sit CHP. The impact of exercise interventions concerning executive functions of children and adolescents with attention-deficit/hyperactive disorder: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2021 May 22;18(1):68. doi: 10.1186/s12966-021-01135-6. PMID 34022908